CLINICAL TRIAL: NCT02181140
Title: Prospective Evaluation of the Significance of the Pro-core® Needle in Differential Diagnosis of Tumorous and Inflammatory Processes
Brief Title: Core Biopsy Endo Sonography Study Evaluation of the Significance of the Pro-core® Needle
Acronym: COS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Medical Director, Interdisciplinary Endoscopy Department and Clinic, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PV 3835
Record Dates: First submitted 2013-07-08; First posted 2014-07-03 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Neoplasm
Keywords: fine needle aspiration; core biopsy; endoscopic ultrasound; space occupying process mediastinal, perigastral, perihilar; suspect lymph nodes mediastinal, perigastral or perihilar; diagnostic accuracy of EUS guided core biopsy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS guided FNA and fine needle punction (Other): punction of endosonographically identified space-occupying process with aspirating fine needle and pro core fine needle in a randomized order
  Interventions: Device: EUS guided FNA and fine needle punction

INTERVENTIONS:
Device: EUS guided FNA and fine needle punction — punction of a suspect area by a EUS guided fine needle as well as pro core fine needle to evacuate histology and smear biologics

SUMMARY:
The study is designed to evaluate the diagnostic accuracy of a new designed endoscopic ultrasonography (EUS) Core biopsy aspiration needle in comparison to a conventional EUS aspiration needle in GI-tumors.

DETAILED DESCRIPTION:
Endoscopic ultrasound is an established examination method for tumors of the gastrointestinal tract and the pancreas. Since imaging by itself is limited in differential diagnosis of tumors, EUS guided fine needle aspiration is seen as a valid complementary method. Since fine-needle aspiration (FNA) is mainly based on cytological diagnostics, this method is limited also because of lacking supplementary immune- histochemical diagnostics. Here, the obtainment of little histologically evaluable tissue samples (punched barrels) would be of benefit.

A new punch needle device called Pro-core needle (Cook)(22 / 19 gauges) offers the possibility of increasing numbers of valid extractions of histologically evaluable tissues due to a better targeted precision and maneuverability in comparison to other devices of that kind (tru-cut needles, e.g.). A little notch at the pinpoint allows the obtainment of little tissue samples, that will be kept within the device by aspiration.

This study compares the obtainment of tissue by Proc-core needle and conventional aspiration punction systems.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for endoscopic ultrasound diagnostics with fine needle biopsies
* age greater than 18 years

Exclusion Criteria:

* difficult or impossible approach to desired structures due to anatomy (postoperative anatomy, e.g.)
* cystic lesion, e.g. cystic pancreas tumors
* coagulopathy
* severe general condition of the patient
* other contraindications for endoscopical ultrasound aided fine needle punction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — University Hospital Eppendorf, Hamburg
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Parikh P, Shiloach M, Cohen ME, Bilimoria KY, Ko CY, Hall BL, Pitt HA. Pancreatectomy risk calculator: an ACS-NSQIP resource. HPB (Oxford). 2010 Sep;12(7):488-97. doi: 10.1111/j.1477-2574.2010.00216.x. PMID 20815858
- [Background] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702
- [Background] Moller K, Papanikolaou IS, Toermer T, Delicha EM, Sarbia M, Schenck U, Koch M, Al-Abadi H, Meining A, Schmidt H, Schulz HJ, Wiedenmann B, Rosch T. EUS-guided FNA of solid pancreatic masses: high yield of 2 passes with combined histologic-cytologic analysis. Gastrointest Endosc. 2009 Jul;70(1):60-9. doi: 10.1016/j.gie.2008.10.008. Epub 2009 Apr 25. PMID 19394012
- [Background] Takahashi K, Yamao K, Okubo K, Sawaki A, Mizuno N, Ashida R, Koshikawa T, Ueyama Y, Kasugai K, Hase S, Kakumu S. Differential diagnosis of pancreatic cancer and focal pancreatitis by using EUS-guided FNA. Gastrointest Endosc. 2005 Jan;61(1):76-9. doi: 10.1016/s0016-5107(04)02224-2. PMID 15672060
- [Background] Iglesias-Garcia J, Dominguez-Munoz E, Lozano-Leon A, Abdulkader I, Larino-Noia J, Antunez J, Forteza J. Impact of endoscopic ultrasound-guided fine needle biopsy for diagnosis of pancreatic masses. World J Gastroenterol. 2007 Jan 14;13(2):289-93. doi: 10.3748/wjg.v13.i2.289. PMID 17226911
- [Background] Sudhoff T, Hollerbach S, Wilhelms I, Willert J, Reiser M, Topalidis T, Schmiegel W, Graeven U. [Clinical utility of EUS-FNA in upper gastrointestinal and mediastinal disease]. Dtsch Med Wochenschr. 2004 Oct 15;129(42):2227-32. doi: 10.1055/s-2004-831867. German. PMID 15483756
- [Background] Aithal GP, Anagnostopoulos GK, Tam W, Dean J, Zaitoun A, Kocjan G, Ragunath K, Pereira SP. EUS-guided tissue sampling: comparison of "dual sampling" (Trucut biopsy plus FNA) with "sequential sampling" (Trucut biopsy and then FNA as required). Endoscopy. 2007 Aug;39(8):725-30. doi: 10.1055/s-2007-966400. Epub 2007 Jul 10. PMID 17620230
- [Background] Wittmann J, Kocjan G, Sgouros SN, Deheragoda M, Pereira SP. Endoscopic ultrasound-guided tissue sampling by combined fine needle aspiration and trucut needle biopsy: a prospective study. Cytopathology. 2006 Feb;17(1):27-33. doi: 10.1111/j.1365-2303.2006.00313.x. PMID 16417562
- [Background] Shah SM, Ribeiro A, Levi J, Jorda M, Rocha-Lima C, Sleeman D, Hamilton-Nelson K, Ganjei-Azar P, Barkin J. EUS-guided fine needle aspiration with and without trucut biopsy of pancreatic masses. JOP. 2008 Jul 10;9(4):422-30. PMID 18648133
- [Background] Storch I, Shah M, Thurer R, Donna E, Ribeiro A. Endoscopic ultrasound-guided fine-needle aspiration and Trucut biopsy in thoracic lesions: when tissue is the issue. Surg Endosc. 2008 Jan;22(1):86-90. doi: 10.1007/s00464-007-9374-x. Epub 2007 May 4. PMID 17479313
- [Background] Storch I, Jorda M, Thurer R, Raez L, Rocha-Lima C, Vernon S, Ribeiro A. Advantage of EUS Trucut biopsy combined with fine-needle aspiration without immediate on-site cytopathologic examination. Gastrointest Endosc. 2006 Oct;64(4):505-11. doi: 10.1016/j.gie.2006.02.056. Epub 2006 Jun 6. PMID 16996340
- [Background] Saftoiu A, Vilmann P, Guldhammer Skov B, Georgescu CV. Endoscopic ultrasound (EUS)-guided Trucut biopsy adds significant information to EUS-guided fine-needle aspiration in selected patients: a prospective study. Scand J Gastroenterol. 2007 Jan;42(1):117-25. doi: 10.1080/00365520600789800. PMID 17190771
- [Background] Sakamoto H, Kitano M, Komaki T, Noda K, Chikugo T, Dote K, Takeyama Y, Das K, Yamao K, Kudo M. Prospective comparative study of the EUS guided 25-gauge FNA needle with the 19-gauge Trucut needle and 22-gauge FNA needle in patients with solid pancreatic masses. J Gastroenterol Hepatol. 2009 Mar;24(3):384-90. doi: 10.1111/j.1440-1746.2008.05636.x. Epub 2008 Nov 20. PMID 19032453
- [Background] Siddiqui UD, Rossi F, Rosenthal LS, Padda MS, Murali-Dharan V, Aslanian HR. EUS-guided FNA of solid pancreatic masses: a prospective, randomized trial comparing 22-gauge and 25-gauge needles. Gastrointest Endosc. 2009 Dec;70(6):1093-7. doi: 10.1016/j.gie.2009.05.037. Epub 2009 Jul 28. PMID 19640524
- [Background] Jenssen C, Faiss S, Nurnberg D. [Complications of endoscopic ultrasound and endoscopic ultrasound-guided interventions - results of a survey among German centers]. Z Gastroenterol. 2008 Oct;46(10):1177-84. doi: 10.1055/s-2008-1027334. Epub 2008 Oct 20. German. PMID 18937186
- [Background] Bournet B, Migueres I, Delacroix M, Vigouroux D, Bornet JL, Escourrou J, Buscail L. Early morbidity of endoscopic ultrasound: 13 years' experience at a referral center. Endoscopy. 2006 Apr;38(4):349-54. doi: 10.1055/s-2005-921173. PMID 16680633
- [Background] Mortensen MB, Fristrup C, Holm FS, Pless T, Durup J, Ainsworth AP, Nielsen HO, Hovendal C. Prospective evaluation of patient tolerability, satisfaction with patient information, and complications in endoscopic ultrasonography. Endoscopy. 2005 Feb;37(2):146-53. doi: 10.1055/s-2005-861142. PMID 15692930
- [Background] Al-Haddad M, Wallace MB, Woodward TA, Gross SA, Hodgens CM, Toton RD, Raimondo M. The safety of fine-needle aspiration guided by endoscopic ultrasound: a prospective study. Endoscopy. 2008 Mar;40(3):204-8. doi: 10.1055/s-2007-995336. Epub 2007 Dec 4. PMID 18058615
- [Background] Williams DB, Sahai AV, Aabakken L, Penman ID, van Velse A, Webb J, Wilson M, Hoffman BJ, Hawes RH. Endoscopic ultrasound guided fine needle aspiration biopsy: a large single centre experience. Gut. 1999 May;44(5):720-6. doi: 10.1136/gut.44.5.720. PMID 10205212
- [Background] O'Toole D, Palazzo L, Arotcarena R, Dancour A, Aubert A, Hammel P, Amaris J, Ruszniewski P. Assessment of complications of EUS-guided fine-needle aspiration. Gastrointest Endosc. 2001 Apr;53(4):470-4. doi: 10.1067/mge.2001.112839. PMID 11275888
- [Background] Wiersema MJ, Vilmann P, Giovannini M, Chang KJ, Wiersema LM. Endosonography-guided fine-needle aspiration biopsy: diagnostic accuracy and complication assessment. Gastroenterology. 1997 Apr;112(4):1087-95. doi: 10.1016/s0016-5085(97)70164-1. PMID 9097990
- [Background] Buscarini E, De Angelis C, Arcidiacono PG, Rocca R, Lupinacci G, Manta R, Carucci P, Repici A, Carrara S, Vallisa D, Buscarini L, Cosentino F, Pera A, Rizzetto M, Testoni PA, Zambelli A. Multicentre retrospective study on endoscopic ultrasound complications. Dig Liver Dis. 2006 Oct;38(10):762-7. doi: 10.1016/j.dld.2006.06.005. Epub 2006 Jul 13. PMID 16843076
- [Result] Sterlacci W, Sioulas AD, Veits L, Gonullu P, Schachschal G, Groth S, Anders M, Kontos CK, Topalidis T, Hinsch A, Vieth M, Rosch T, Denzer UW. 22-gauge core vs 22-gauge aspiration needle for endoscopic ultrasound-guided sampling of abdominal masses. World J Gastroenterol. 2016 Oct 21;22(39):8820-8830. doi: 10.3748/wjg.v22.i39.8820. PMID 27818598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EUS Guided FNA and Fine Needle Punction
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EUS Guided FNA and Fine Needle Punction
Number analyzed (Participants) | 56
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 29
Region of Enrollment [Number; unit: participants]
  Germany | 56

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy of Pro-core needle (22 G) will be compared to conventional fine needle aspiration (22 G). Therefore EUS-FNA with both needles is undertaken in a random order in each lesion. For Pro-core needle, a histological / cytological diagnosis and quality assessment will be made by pathologists.For Echotip aspiration needle, reference cytology evaluation is done by cytology experts.
  The histopathological diagnosis after surgery or the clinical follow up of at least one year after EUS FNA is current standard.
Time Frame: up to 1 year
Measure: Number; unit: Diagnostic accuracy (%)
Groups:
- EUS Guided Pro Core FNA: EUS guided punction of a lesion by pro core fine needle to evacuate histology and smear biologics
Arm/Group | EUS Guided Pro Core FNA
Number analyzed (Participants) | 56
Diagnostic accuracy (%) | 84

2. Secondary Outcome: EUS Pro Core FNA: Histology Samples
Description: Histology (not cytology) samples for Pro-core Needle: Number of adequately evaluable histology samples
Time Frame: day 0 and day 14
Population: Histology (not cytology) samples for Pro-core Needle
Measure: Number; unit: participants
Groups:
- EUS Guided Pro Core FNA: EUS guided Pro core FNA: Histology samples (not cytology)
Arm/Group | EUS Guided Pro Core FNA
Number analyzed (Participants) | 56
participants | 36

3. Secondary Outcome: Complication Rates
Description: Complication rates of EUS FNA
Time Frame: day 0 and day 14
Measure: Number; unit: participants
Groups:
- EUS Guided FNA: EUS FNA of lesions with aspirating fine needle and pro core fine needle in a randomized order
Arm/Group | EUS Guided FNA
Number analyzed (Participants) | 56
participants | 0

ADVERSE EVENTS:
Time Frame: 1 fortnight
Arm/Group | EUS Guided FNA
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No